CLINICAL TRIAL: NCT06692335
Title: A Randomized Controlled Trial of High-Intensity Focused Ultrasound (HIFU) Versus Myomectomy for the Treatment of Symptomatic Uterine Fibroids
Brief Title: HIFU Versus Myomectomy for the Treatment of Symptomatic Uterine Fibroids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SYMPHOROSA SHING CHEE, Consultant and Honorary Clinical Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2024.176
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Uterine Fibroids (UF)
Keywords: symptomatic uterine fibroid; Menorrhagia; Dysmenorrhea
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Dysmenorrhea | interventions — Uterine Myomectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU group (Active Comparator): All women in the HIFU group will undergo pelvic MRI scans, including T1- and T2-weighted imaging, for fibroid localization and treatment planning. The HIFU treatment will utilize the Haifu JC 200 system under real-time ultrasound guidance, with participants positioned prone in a water-filled generator chamber. Conscious sedation will be administered using fentanyl and midazolam, adjusted based on pain tolerance. Acoustic output power will range from 300 to 400W, with treatment energy tailored to participant feedback and ultrasound imaging.
  Post-procedure, participants will be monitored for 4-6 hours, with discharge criteria including dietary tolerance and urination. Data on pain, skin condition, and adverse events will be collected.
  Before discharge, participants will complete a Client Satisfaction questionnaire and will receive analgesics, along with instructions to document menstrual cycles using the PBAC chart.
  Interventions: Procedure: High-Intensity Focused Ultrasound (HIFU)
- Myomectomy group (Placebo Comparator): Myomectomy will be performed using laparoscopic, open, or hysteroscopic techniques by accredited HKCOG gynecologists.
  Key metrics such as blood loss, intraoperative and postoperative complications, whether the endometrial cavity was entered, length of hospital stay, need for blood transfusion, and readmissions will be meticulously recorded. A complete blood count will be assessed approximately 6 hours post-surgery. Patients will be monitored for blood pressure and pulse per departmental protocol.
  Typically, those undergoing hysteroscopic myomectomy are discharged the same day, while laparoscopic or open myomectomy patients are discharged within 1 to 3 days.
  Before discharge, women will complete a Client Satisfaction questionnaire and will receive analgesics, along with instructions to document their menstrual cycle, flow, and dysmenorrhea using the PBAC chart.
  Interventions: Procedure: myomectomy

INTERVENTIONS:
Procedure: High-Intensity Focused Ultrasound (HIFU) — The HIFU treatment will utilize the Haifu JC 200 system under real-time ultrasound guidance, with participants positioned prone in a water-filled generator chamber. Conscious sedation will be administered using fentanyl and midazolam, adjusted based on pain tolerance. Acoustic output power will range from 300 to 400W.
  Arms: HIFU group
Procedure: myomectomy — Laparoscopic or open or hysteroscopic myomectomy will be performed.
  Arms: Myomectomy group

SUMMARY:
The goal of this clinical trial is to learn if High-Intensity Focused Ultrasound (HIFU) is as effective as myomectomy for treating symptomatic uterine fibroids in women aged 18 to 50. The main questions it aims to answer are:

Is HIFU as effective as myomectomy in improving quality of life for women with uterine fibroids? How do the recovery times and complications compare between HIFU and myomectomy? Researchers will compare the outcomes of women receiving HIFU treatment to those undergoing myomectomy to see if HIFU offers similar or better results with fewer complications.

Participants will:

Undergo an initial medical assessment, including ultrasounds and blood tests. Receive either HIFU treatment or myomectomy based on random assignment. Complete questionnaires about their symptoms and quality of life before treatment and at follow-up visits (3 and 6 months post-treatment).

Be monitored for any complications and recovery progress during follow-up.

DETAILED DESCRIPTION:
This multicenter, randomized controlled trial (RCT) aims to compare the effectiveness, safety, and quality of life impacts between HIFU and myomectomy in treating symptomatic uterine fibroids. The study will adhere to the International Council for Harmonisation's Good Clinical Practice (ICH-GCP) guidelines and the Declaration of Helsinki.

Recruitment and Baseline Characteristics:

Women aged 18 to 50 who present with symptomatic uterine fibroids will be recruited from gynecology clinics within the New Territories East Cluster (NTEC) and Kowloon East Cluster (KEC). The recruitment process will involve a thorough review of participants' gynecological and medical histories, physical examinations, blood tests and imaging studies to assess fibroid characteristics.

All participants will be invited to fill in the Chinese validated Uterine Fibroid Symptom and Health-related Quality of Life questionnaire (UFS-QOL), Short Form-12 questionnaire (SF-12); and Pictorial Blood loss Assessment Chart (PBAC) to document menstrual cycles and any dysmenorrhea experienced.

Randomization:

Participants meeting the inclusion criteria will be consented and randomized in a 1:1 ratio to either the HIFU group or the myomectomy group via permuted-block randomization. Randomization will be conducted by a research assistant using sealed, opaque envelopes containing computer-generated treatment assignments.

Interventions:

HIFU Protocol:

Pre-Treatment Imaging: All participants in the HIFU group will undergo a pelvic MRI for localization and assessment of fibroids.

HIFU Treatment:

The Haifu JC 200 Focused Ultrasound Tumor Therapeutic System will be employed. Participants will lie in a prone position with their lower abdomen submerged in degassed water. Conscious sedation will be achieved using fentanyl and midazolam, adjusted per participant feedback during the procedure.

Postoperative Care and Discharge Planning:

After treatment, patients will be observed for 4-6 hours in the ward for any immediate side effects, with discharge criteria based on their ability to tolerate food and mobilize.

Myomectomy Surgical Approach:

Myomectomy will be conducted using laparoscopic, open, or hysteroscopic techniques.

Intraoperative Monitoring:

Key metrics such as blood loss, complications, and whether the endometrial cavity is entered will be meticulously recorded.

Postoperative Care and Discharge Planning:

Patients will be monitored according to the department's protocol, with blood tests performed at approximately 6 hours post-surgery to evaluate hemoglobin levels. Similar to the HIFU group, women will be discharged with analgesics and instructed to document their menstrual symptoms.

Post-Procedure Documentation:

Baseline characteristics, pain levels, skin condition, neurological symptoms, and other adverse events will be documented. All participants will be asked to fill in the Client Satisfaction Questionnaire (CSQ-8) and PBAC.

Follow-Up Procedures:

All participants will be followed up by a telephone interview at 2 weeks, and a face-to-face assessment at 3 months and 6 months post-treatment. During these clinical visits, vital signs will be monitored, and participants will complete the UFS-QOL, SF-12, and CSQ-8. Investigators blinded to group assignments will perform physical assessments and ultrasound scans to evaluate uterine size and fibroid volume.

Data Processing and Analysis:

Data analysis will be conducted using SPSS 29.0. An intention-to-treat approach will be employed. Categorical data will be analyzed using Chi-square or Fisher exact tests. Continuous variables will be assessed using appropriate t-tests or non-parametric equivalents. Both univariate and multivariate analyses will be used to identify factors associated with treatment outcomes.

Hypothesis:

The findings from this RCT could significantly impact clinical practice by offering a less invasive treatment alternative for women with symptomatic uterine fibroids, potentially leading to improved quality of life and fertility preservation. The study's comprehensive design and rigorous methodology aim to address existing gaps in the literature regarding the effectiveness and safety of HIFU compared to traditional surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 50 years-old
* Pre or peri menopausal with FSH less than 25 mIU/ml
* BMI < 33 kg/m2 or abdominal wall thickness < 5 cm
* Uterine size ≤18 weeks based on physical exam assessment
* Dominant intramural fibroid ≥ 3cm and ≤ 10cm on imaging
* Symptomatic fibroids cause menorrhagia, pressure, or pelvic pain
* Willing and able to give informed consent

Exclusion Criteria:

* Patient with other pelvic mass indicated by history or magnetic resonance imaging (MRI) such as endometriosis, abnormal adnexal mass, ovarian tumor, acute or chronic pelvic inflammatory disease
* Morbid obesity
* Inability to lie in a prone position for more than 2 hours
* Extensive abdominal scar on the acoustic channel
* Women with pregnancy, lactation or menopause
* Uterine premalignant or malignant pathologies or pathology other than uterine fibroid cannot be ruled out through detailed clinical assessment and investigation including MRI
* Rapid growth of fibroids, defined as a doubling in size in 6 months
* History of or current thromboembolic event (deep vein thrombosis, pulmonary embolus, stroke)
* Coagulation problem or using medication which affect clotting function
* History of pelvic irradiation
* Pedunculated submucosal or subserosal fibroid of size ≧5cm and with a stalk less than 25% of the maximal fibroid diameter
* Cervical/ broad ligament fibroid
* Contraindication to MRI due to severe claustrophobia or implanted metallic device.
* Co-existing adenomyosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of quality of life by Uterine Fibroid Symptom health-related Quality of Life questionnaire (UFS-QOL) from baseline to 3 months after HIFU or myomectomy | From enrollment to the end of treatment at 3 months
  The efficacy of treatment using the Uterine Fibroid Symptom health-related Quality of Life questionnaire (UFS-QOL), changes from baseline to 3 months post-treatment
Change of quality of life by Uterine Fibroid Symptom health-related Quality of Life questionnaire (UFS-QOL) from baseline to 6 months after HIFU or myomectomy | From enrolment to the end of treatment at 6 months
  The efficacy of treatment using the Uterine Fibroid Symptom health-related Quality of Life questionnaire (UFS-QOL), changes from baseline to 6 months post-treatment

SECONDARY OUTCOMES:
Change of health-related quality of life by Short Form-12 questionnaire (SF-12) from baseline to 3 months after HIFU or myomectomy | From enrolment to the end of treatment at 3 months
  The efficacy of treatment in health-related quality of life by Short Form-12 questionnaire (SF-12), changes from baseline to 3 months
Change of health-related quality of life by Short Form-12 questionnaire (SF-12) from baseline to 6 months after HIFU or myomectomy | From enrolment to the end of treatment at 6 months
  The efficacy of treatment in health-related quality of life by Short Form-12 questionnaire (SF-12), changes from baseline to 6 months
Change of Pictorial Blood loss Assessment Chart (PBAC) score from baseline to 3 months after HIFU or myomectomy | From enrolment to the end of treatment at 3 months
  The efficacy of treatment in PBAC score, changes from baseline to 3 months post-treatment
Change of Pictorial Blood loss Assessment Chart (PBAC) score from baseline to 6 months after HIFU or myomectomy | From enrolment to the end of treatment at 6 months
  The efficacy of treatment in PBAC score, changes from baseline to 6 months post-treatment
Change of scores by Client Satisfaction questionnaire (CSQ-8) from baseline to 3 months after HIFU or myomectomy | From enrolment to the end of treatment at 3 months
  The efficacy of treatment in satisfaction score by Client Satisfaction questionnaire (CSQ-8), changes from baseline to 3 months
Change of scores by Client Satisfaction questionnaire (CSQ-8) from baseline to 6 months after HIFU or myomectomy | From enrolment to the end of treatment at 6 months
  The efficacy of treatment in satisfaction score by Client Satisfaction questionnaire (CSQ-8), changes from baseline to 6 months
Change of haemoglobin from baseline to 3 months after HIFU or myomectomy | From enrolment to the end of treatment at 3 months
  The efficacy of treatment in haemoglobin, changes from baseline to 3 months post-treatment
Change of haemoglobin from baseline to 6 months after HIFU or myomectomy | From enrolment to the end of treatment at 6 months
  The efficacy of treatment in haemoglobin, changes from baseline to 6 months post-treatment
Change of fibroid volume from baseline to 3 months after HIFU or myomectomy | From enrolment to the end of treatment at 3 months
  The efficacy of treatment in fibroid volume, changes from baseline to 3 months post-treatment
Change of fibroid volume from baseline to 6 months after HIFU or myomectomy | From enrolment to the end of treatment at 6 months
  The efficacy of treatment in fibroid volume, changes from baseline to 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shing Chee Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
We have not mentioned data-sharing in protocol and approved by ethics committee.